## STU#:00204116 NCT # NCT03316118

# STATISTICAL ANALYSIS PLAN Version date 09/12/2017

### PROTOCOL TITLE:

A Comparison of Analgesic Efficacy of Ultrasound-Guided Genicular Nerve Block versus Saline Injection for Total Knee Replacement: a Prospective, Randomized Controlled Trial

#### PRINCIPAL INVESTIGATOR:

Antoun Nader, MD

Institution: Northwestern University, Feinberg School of Medicine

Department: Anesthesiology

Address: 251 East Huron Street, Feinberg Pavilion 5-704, Chicago, IL 60611

Email Address: anader2@northwestern.edu

Phone: (312) 695-3045 Fax: (312) 695-5876

#### STU00204116

#### **Statistical Plan**

Pain burden defined as the area under the numeric rating score for pain for the first 36 hours will be calculated using the trapezoidal method. Time to report first pain and overall patient satisfaction between groups will be compared using the Kruskal-Wallis H test.